CLINICAL TRIAL: NCT06952972
Title: MorphECOS - Evaluation of the Influence of Fatigue and Sleep on the Performance of 2nd Cycle Medical Students (OSCE): a Single-centre Observational Study
Brief Title: MorphECOS - Evaluation of the Influence of Fatigue and Sleep on the Performance of 2nd Cycle Medical Students (OSCE)
Acronym: MorphECOS
Status: Completed | Type: Observational
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, Evan GOUY, Principal Investigator, Claude Bernard University
Other Study IDs: MorphECOS
Record Dates: First submitted 2025-02-03; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Fatigue Intensity; Sleep; Sleep Deprivation; Circadian Rhythm
MeSH Terms: conditions — Fatigue; Sleep Deprivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 5th year of medical curriculum: 5th year of medical curriculum
- 6th year of medical curriculum: 6th year of medical curriculum

SUMMARY:
Objective and Structured Clinical Examinations (OSCEs) has been incorporated recently in the certification process as a final national undergraduate ranking examination. This exam is a challenge for medical students.

The aim of this study is to better characterise the population of students taking the OSCEs on the subject of sleep and fatigue and to assess whether these factors have an impact on their performance in the OSCEs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of legal age, enrolled in the 2nd cycle médical program at the Lyon Est Faculty of Medicine (Claude Bernard Lyon 1 University), taking part in the annual session (February or March 2025) of the faculty's OSCEs and having agreed to participate by completing and signing the dedicated written consent form.

Exclusion Criteria:

* abstenteism or Premature end to the OSCE session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 2nd cycle médical program
Sampling Method: Non-Probability Sample
Enrollment: 619 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
PERFORMANCE | obtained seven days after the objectif structured clinical examination
  Score at the objectif structured clinical examination exam from 0 minimum to 200 points maximum

SECONDARY OUTCOMES:
Significant difference in student performance per station and per item | obtained seven days after the objectif structured clinical examination
  Significant difference in student performance per station and per item
Significant difference in Visual Analog Scale response according to the different profiles | Two times : 1 hour before and 1 hour after the OSCE session
  Significant difference in Visual Analog Scale response according to the different profiles

CONTACTS AND LOCATIONS:
Locations (1):
- Claude Bernard University, Lyon, France, France

IPD SHARING:
Plan to Share IPD: No
Not provided for in the protocol.